CLINICAL TRIAL: NCT04837105
Title: Serious Game-based Intervention in Gait Rehabilitation for Children With Cerebral Palsy: Randomized Control Trial
Brief Title: Serious Game-based Intervention in Gait Rehabilitation for Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ellen Poidatz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARROW CP
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy; Gait Disorders, Neurologic
Keywords: physiotherapy; gait rehabilitation; serious game; multi level surgery
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: randomized control trial - 2 groups
Who Masked: Outcomes Assessor
Masking Description: Pre-test and post-test evaluation are made by one physiotherapist ignoring the patient's arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Classic rehab (physio including strength rehab, fitness, motor activity...) + treadmill gait training 3*/week/4weeks:
  5 minutes of warm-up with gradual increase in treadmill speed, max 20 minutes of walking at 80% of maximum speed, 5 minutes of active recovery with gradual decrease in treadmill speed.
  (protocol from Grecco et al.)
  Interventions: Other: Treadmill
- Test group (Experimental): Classic rehab - same as control group - (physio including strength rehab, fitness, motor activity...) + overground ARROW CP gait training 3*/week/4weeks:
  walking sprint session at maximal speed with gradual increase in number of repetitions over the weeks.
  (protocol from Verschuren et al.)
  Interventions: Other: Serious game ARROW CP

INTERVENTIONS:
Other: Serious game ARROW CP — ARROW CP is developed for Microsoft Hololens headset. Feedback on gait performance are delivering to the participant in real time and with delay. Participants have to walk at their maximal speed during "sprint session".
  Arms: Test group
Other: Treadmill — Participant walk on a treadmill at 80% of their maximal speed during maximum 20 minutes (+5 min warm-up / 5 min cool-down)
  Arms: Control group

SUMMARY:
Cerebral palsy (CP) is defined as a group of movement and posture disorders that cause activity limitation due to brain damage during fetal development or in the first year of life. Motor activities, and in particular walking, can be affected by many factors including sensory deficits, biomechanical and postural limitations, muscle weakness and spasticity. Theories of gait training guide rehabilitation management strategies. Among these, intensification, variability and specific training of walking parameters (speed, step length, cadence) have shown their effectiveness. Delivering sensory feedback during gait rehabilitation exercises is a complementary approach to improve motor learning during rehabilitation. On the other hand, motivation is a key factor in the success of rehabilitation. The addition of walking exercises performed through a serious game in augmented reality (AR) appears relevant for the rehabilitation of children with CP after surgery.

The serious game ARRoW-CP is based on the latest advances in the literature in terms of gait rehabilitation protocol but also on the results of a clinical study conducted by our team, to identify the best feedback modalities to be delivered during the serious rehabilitation game.

DETAILED DESCRIPTION:
This study is a randomized control trial.

Participants are children with cerebral palsy having a single event multi level surgery. They are involving in a rehabilitation protocol in the same rehab center.

Two groups are formed:

* control group: classic rehab+children have treadmill gait protocol during 4 weeks
* test group : classic rehab+children have gait training with the ARROW CP serious game.

ARROW CP game is developed for augmented reality headset (Microsoft Hololens). It delivers feedback in real time and with delay on participant gait performance. This game has been developed by researchers (Fondation Ellen Poidatz, France).

The aims of this study are:

1. . To determine the impact on spatiotemporal gait parameters of intensive gait rehabilitation involving the use of a serious AR game in children and adolescents with cerebral palsy.
2. To explore the effects of playing a serious game on functional abilities
3. To assess motivation, satisfaction and adherence to treatment

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of CP mentioned in the medical record
* Minor child for the entire duration of the protocol, i.e. between 10 and 17 years of age (the child must be less than 18 years of age at the time of the last check-up scheduled 1 year after inclusion in the study)
* Global Motor Function Classification System (GMFCS) levels I to III
* Functional Mobility Scale 50 meters rating superior or equal to 2 (ability to walk on 50m using a walker or frame without help from another person)
* Ability to cooperate, understand and follow simple instructions to play.
* Patient affiliated to the French social security system
* Voluntary patient whose parents have given their consent for their child to participate in the study
* Patient who has undergone multisite surgery of the lower limbs including bone procedures at least 7 weeks before the start of the procedure

Exclusion Criteria:

* A diagnosis of photosensitive epilepsy mentioned in the medical file AND/OR a mention in the child's medical file or by the parents or by the child of a history of epileptic seizures occurring during the practice of a video game
* A visual, cognitive or auditory impairment at a level that would interfere with playing the game. The patient must have normal or corrected vision and hearing.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
6 minutes walking test | 6 minutes
  Aim of the measurement: To quantify changes in the parameters of walking quality (speed, cadence, step length).
  Procedure: The patient is instructed to walk for 6 minutes in an unobstructed corridor. The distance walked is recorded for the calculation of walking speed. Fatigue is assessed with a Borg scale and heart rate is continuously recorded.

SECONDARY OUTCOMES:
Muscle power sprint test | 10 minutes
  Aim of the measurement: To assess the anaerobic capacity of children with motor disabilities.
  Procedure: The patient is asked to perform six 15-metre walking sprints, with 10 seconds of rest between each sprint. The average and maximum power are calculated based on the speeds achieved during the sprints.
Shuttle run test I and II (adapted for children with CP) | 20 minutes
  In this test, the child must walk between 2 poles spaced 10 metres apart following the "beep rhythm" imposed by a pre-recorded soundtrack. The soundtrack includes an increase in walking speed of 0.25 km/h every minute.
  (Verschuren et al.)
Questionnaire (PACES) | 10 minutes
  To assess enjoyment for both control and test group, the 16-items of the Physical Activity Enjoyment Scale (PACES) will be used. The PACES is a valid and re- liable measure of physical activity enjoyment. It has been used in many studies assessing the effectiveness of VR therapy This questionnaire will be presented to the participant at the end of the last session.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ellen Poidatz, Saint-Fargeau-Ponthierry, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guinet AL, Bams M, Payan-Terral S, Khouri N, Otmane S, Bouyer G, Desailly E. Effect of an augmented reality active video game for gait training in children with cerebral palsy following single-event multilevel surgery: protocol for a randomised controlled trial. BMJ Open. 2022 Oct 10;12(10):e061580. doi: 10.1136/bmjopen-2022-061580. PMID 36216413
- See also: Fondation Ellen Poidatz ARROW CP — https://www.fondationpoidatz.com/arrow-cp/